CLINICAL TRIAL: NCT00110786
Title: A Double Blind Study to Investigate the Clinical Efficacy and Safety of Ragweed MATAMPL (Allergy Therapeutics®), Pollinex®-R (Allergy Therapeutics®) and Placebo in Patients With Seasonal Allergic Rhinitis With Ragweed Allergy, in an Environmental Exposure Chamber (EEC) Model, With Follow-Up During a Natural Ragweed Pollen Season
Brief Title: Investigation of Efficacy and Safety of Ragweed MATAMPL, Pollinex-R and Placebo in Patients With Ragweed Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RagweedMATAMPL204; P2DP05001
Record Dates: First submitted 2005-05-13; First posted 2005-05-16 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2009-09

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy; Ragweed; Environmental Exposure Chamber
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: Ragweed MATAMPL

SUMMARY:
Ragweed MATAMPL has been developed to provide pre-seasonal specific immunotherapy for patients with hypersensitivity to ragweed pollen (hay fever). This novel formulation is designed to provide a vaccine that will be efficacious with only four escalating dose injections administered before the start of the pollen season.

In this study, the safety and efficacy of Ragweed MATAMPL will be assessed by exposing allergic subjects to Ragweed pollen in an environmental exposure chamber (EEC). Patient symptomatic response to pollen and patient quality of life in the EEC will be determined.

DETAILED DESCRIPTION:
Allergic rhinitis is a nasal inflammatory disorder initiated by an immunoglobulin-E (IgE) mediated hypersensitivity to allergens. This condition is characterized by sneezing, rhinorrhea, nasal itching and congestion. When a patient is exposed to an allergen to which they are sensitive, the allergen cross-links with the Ig E antibody, which is bound to the surface of tissue mast cells. This cross-linking then triggers the release of proinflammatory substances, such as histamine and eicosanoids, and is known as the early response. In a skin prick test, this reaction produces a wheal-and-flare response. Normally, systemic exposure to an allergen also leads to the more prolonged late reaction, in which eosinophils, basophils, and activated T cells are recruited to the site of exposure. The recruited T cells also secrete inflammatory cytokines, such as interleukin-4 (IL-4) and IL-5, typically associated with helper T cells type 2 (TH2), which further propagate the inflammatory cascade. Typically, the early response occurs within 15 to 30 minutes (but as quickly as a few seconds) and usually resolves within 1 to 3 hours, and the late response occurs within 6 to 12 hours and resolves in 24 hours.

Allergic vaccination (AV), also referred to as immunotherapy or allergen-specific immunotherapy (SIT), is a curative approach that is available for allergic diseases, which directly treats the underlying disease. AV is the practice of administering gradually increasing quantities of an allergen extract to an allergic patient to ameliorate the symptoms associated with the subsequent exposure to the causative allergen. AV is believed to exert its beneficial effects on the immune system, at least in part, by modifying the T-lymphocyte response to subsequent natural allergen exposure. AV has been shown to inhibit both early and late responses to allergen exposure. AV acts on T cells to modify peripheral and mucosal TH2 responses to allergen in favor of helper T cell type 1 (TH1) responses. One of the hallmarks of successful AV is the redressing of a "healthy" TH1/TH2-balance.

Although efficacious, immunotherapy is generally considered a long-term disease modifying measure that requires months to years of treatment, entails multiple injection regimens and involves some risk for adverse immune reactions.

Recent improvements, such as optimal dosing, allergen modification (to reduce allergenicity while maintaining immunogenicity), adjuvant adsorption (to control release) and adjuvant activity (to assist immunomodulatory action) are being explored to reduce the risk of anaphylaxis and decrease the commitment to multiple injections.

A novel allergy vaccine (Ragweed MATAMPL) has been developed for the prevention or relief of allergic symptoms caused by a variety of pollens. Ragweed MATAMPL, which contains the allergens of ragweed (chemically modified by glutaraldehyde) adsorbed onto L-tyrosine with the addition of the adjuvant monophosphoryl lipid A (MPL), is being evaluated for the specific treatment of ragweed seasonally induced allergic rhinitis. Ragweed MATAMPL is intended for use as a pre-seasonal therapeutic allergy vaccine in patients with proven seasonal allergic rhinitis and conjunctivitis due to IgE mediated allergy to ragweed. This novel vaccine formulation is designed to provide a vaccine that will be efficacious with only four escalating dose injections, in contrast to the longer schedules currently in use.

This placebo-controlled clinical trial is designed to evaluate the safety and efficacy of Ragweed MATAMPL as determined by patient symptomatic response to pollen and patient quality of life in an environmental exposure chamber (EEC) that reproduces the clinical setting. The development of the EEC, which delivers a controlled pollen challenge over time and allows evaluation of a patient's response at any time point throughout the challenge process, provides the opportunity to examine various aspects of efficacy of anti-allergic treatments within a single center at various times of the year. The EEC affords a more controlled environment than natural pollen exposure in which variables such as unpredictable pollen levels, varying weather conditions during the study period, and varying levels of pollen exposure within the patient population are eliminated. Furthermore, the question of patient compliance is largely eliminated because the patients are scrutinized closely while they are recording symptoms. In addition, an EEC study is an acceptable study model for determining the dose response for an allergic rhinitis drug as outlined in the draft U.S. Food and Drug Administration (FDA) guidelines "Allergic Rhinitis Clinical Development Programs for Drug Products," April 2000.

ELIGIBILITY:
Inclusion Criteria:

* at least a 2-year clinical history of seasonal allergic rhinitis
* allergy to a ragweed allergen, defined by positive case history and positive skin prick test
* Specific IgE for ragweed as documented by a radioallergosorbent test (RAST), or equivalent test, with class >= 2
* minimum qualifying symptom scores on at least one Symptom Diary Card during EEC exposure at both Visits 4 and 5.
* Patients must observe drug washout times listed in the protocol prior to Screening.
* Males or non-pregnant, non-lactating females who are post-menopausal or naturally or surgically sterile
* Females of childbearing potential should be using acceptable birth control methods
* Patients who are normally active and otherwise judged to be in good health
* Patients must be willing and able to give written informed consent and must provide this consent
* Patients must be willing and able to attend required study visits
* Patients must be able to follow instructions

Exclusion Criteria:

* Symptomatic for allergic rhinitis or allergic conjunctivitis from allergy to grass or trees
* Symptomatic for significant perennial rhinitis
* Concurrent disease that might complicate or interfere with investigation or evaluation of the study medications
* Concurrent use of any prohibited medication(s) or inadequate washout of medication
* Chronic or intermittent use of inhaled, oral, intramuscular, intravenous, or potent or super-potent topical corticosteroids
* Chronic use of long acting antihistamines and other concomitant medications that would affect assessment of the effectiveness of study drug(s)
* Any systemic disorder that could interfere with the evaluation of the study medication(s)
* Upper or lower respiratory infection requiring antibiotics within 14 days of the first Baseline EEC Visit
* Diagnosis of sinusitis within 30 days of the first Baseline EEC Visit
* Any ocular disorder (other than allergic conjunctivitis) which could interfere with the evaluation of the study medication
* Hypersensitivity to the study drug excipients
* active or quiescent tuberculous infection of the respiratory tract, untreated local or systemic fungal or bacterial or systemic viral infections or parasitic or ocular herpes simplex
* nasal septal ulcers, nasal surgery or nasal trauma within 90 days of enrollment
* Clinical history of anaphylaxis
* Patients with contraindications for allergy vaccines
* Clinical history of immunodeficiency, including immunosuppressant therapy
* Patients in whom tyrosine metabolism is disturbed
* Patients with contraindications to adrenaline
* Subject is taking β-blockers
* Current diagnosis of chickenpox or measles
* Clinical history of drug or alcohol abuse that would interfere with the patient's participation in the study
* Clinical history of severe or uncontrolled cardiovascular, hepatic, renal and/or other disease/illness that could be expected to interfere with the study
* Clinical history, or evidence, of nasolacrimal drainage system malfunction
* Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol
* Patient that has received Ragweed MATAMPL in any previous clinical trial
* History of immunotherapy with ragweed pollen extract
* Patient received treatment with preparation containing MPL during the past 12 months
* Participation in any other investigational study within 30 days before entry into this study or concomitantly with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-05; Study Completion 2005-12

PRIMARY OUTCOMES:
Assessment of the clinical efficacy of Ragweed MATAMPL versus placebo in reducing seasonal allergic rhinitis (SAR) symptoms caused by ragweed pollen in an Environmental Exposure Chamber (EEC) Model

SECONDARY OUTCOMES:
Comparison of the efficacy of Pollinex-R (modified Ragweed Tyrosine adsorbate) versus placebo in reducing SAR symptoms caused by ragweed pollen in an EEC Model
Assessment of the immunological response to Ragweed MATAMPL, Pollinex-R, versus placebo immunotherapy in patients with SAR
Evaluation of the impact of Ragweed MATAMPL and Pollinex-R versus placebo on quality-of-life in patients with SAR using the Rhinoconjunctivitis Quality of Life Questionnaire for use in the Environmental Exposure Chamber (RQLQ-EEC)
Assessment of the safety and tolerability of Ragweed MATAMPL and Pollinex-R versus placebo in patients with SAR

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International Inc.
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada